CLINICAL TRIAL: NCT01992406
Title: Feasibility, Safety and Outcome of Transrectal Hybrid-NOTES Anterior Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cantonal Hosptal, Baselland (Other)
Responsible Party: Principal Investigator, Daniel Steinemann, MD, Principle Investigator, Cantonal Hosptal, Baselland
Other Study IDs: TRANSRECTAL
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Sigmoid Diverticulosis; Sigmoid Diverticulitis; Colon Adenoma; Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transrectal hybrid-NOTES anterior resection

SUMMARY:
Natural orifice transluminal endoscopic surgery has become an important topic. NOTES access routes give the opportunity to reduce surgical access trauma leading to a more painless surgery and enhancing a fast postoperative recovery. Experience with transvaginal laparoscopic cholecystectomy and transvaginal anterior resection for diverticulitis show that such NOTES procedures are feasible and safe. The complication rate to conventional laparoscopic procedures is similar. Since transvaginal access is impossible in men, an alternative route is missing. There are experimental studies and small case series reporting the feasibility of transrectal anterior resection. However any prospective feasibility study demonstrating the safety of the procedure and functional outcomes (sphincter function) are missing. This study investigates the feasibility, practicability, safety and subjective as well as functional outcome of transrectal hybrid-NOTES anterior resection.

DETAILED DESCRIPTION:
Primary endpoint:

To demonstrate in a prospective cohort study the feasibility (specimen extraction through rectum possible to perform or not), safety (complications graded according to Clavien-Dindo) and postoperative outcome (gastrointestinal quality of life questionnaire and anal sphincter manometry) of routine hybrid-NOTES transrectal anterior resection for benign indication in men and women.

Secondary endpoints:

* quality of life 6 months after surgery
* continence 6 months after surgery
* pain postoperative
* complication rate
* duration of procedure
* lengh of stay

Hypothesis:

The investigators expect specimen extraction through the rectum to be feasible in 80% of cases (in the others an alternative mini-laparotomy has to be performed).

study design: This is an open cohort study on 60 patients. The patients are included before surgery and baseline parameters are put in a registry. There are clinical controls 6 weeks, 3 and 6 months postoperative. 3 and 6 months postoperative as well as preoperative a anorectal manometry is performed.

Inclusion criteria:

- benign indication for left sided colectomy.

exclusion criteria:

* age <18 years
* patient unable to understand informed consent or missing informed consent
* emergency surgery

power calculation: A feasibility of 80% with a precision of 15% is estimated. Given a 5% drop out rate 36 patients are to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* benign indication for left sided colectomy

Exclusion Criteria:

* age below 18 years
* unable to understand informed consent of missing informed consent
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with benign indication for left sided colectomy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Transanal specimen extraction possible or not | at surgery
  Feasibility to remove the specimen (sigmoid colon) through the rectum/anus. If this is not possible during surgery (due to bulky specimen or narrow pelvis) an alternative mini-laparotomy has to be performed.

SECONDARY OUTCOMES:
Number of Participants with postoperative complications (and severity of complications according Clavien-Dindo) | up to 6 weeks postoperative
  Postoperative complications are recorded and graded according to Clavien-Dindo classification. Complication rates and especially occurence of anastomotic leakage and pelvic sepsis will be compared to the literature of current techniques.
continence 6 months postoperative | 6 months postoperative
quality of life | 6 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Zerz, MD, Study Chair — Kantonsspital Baselland, Department of Surgery, Bruderholz
Locations (1):
- Kantonsspital Baselland, Department of Surgery, Bruderholz, Bruderholz, Switzerland

REFERENCES:
- [Derived] Steinemann DC, Zerz A, Germann S, Lamm SH. Anorectal Function and Quality of Life after Transrectal Rigid-Hybrid Natural Orifice Translumenal Endoscopic Sigmoidectomy. J Am Coll Surg. 2016 Aug;223(2):299-307. doi: 10.1016/j.jamcollsurg.2016.04.002. Epub 2016 Apr 13. PMID 27086090